CLINICAL TRIAL: NCT00402818
Title: RESTORE (Raptiva® (Efalizumab) Evaluation of Safety and Treatment Optimization Registry) Observational, Open-label, Multi-centre, Phase IV Study of Subcutaneously Administered Raptiva® (Efalizumab) in the Treatment of Adult Patients With Moderate to Severe Chronic Plaque Psoriasis Who Are Candidates for Treatment With Raptiva®
Brief Title: RESTORE: Raptiva® (Efalizumab) Evaluation of Safety and Treatment Optimization
Acronym: RESTORE
Status: Terminated | Type: Observational
Why Stopped: The study was terminated after the EMEA recommended to suspend the marketing authorisation of Raptiva in the EU
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 26768
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Plaque Psoriasis
Keywords: Moderate to severe plaque psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
RESTORE is an observational, open-label, multi-center, prospective, study enrolling Raptiva® (efalizumab) treated patients with moderate to severe chronic plaque psoriasis. The overall duration of the study is approximately 4 years. Patients will be followed from the time of study enrolment to study/treatment termination; thus active follow-up period will vary across subjects. Raptiva® (efalizumab)treated patients with moderate to severe chronic plaque psoriasis and meeting the inclusion/exclusion criteria specified will be eligible for participation in this study.

Objectives:

* To document and quantify the incidences of adverse events in this patient population
* To explore the association of psoriasis treatments with changes in patient outcomes, quality of life, and treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old.
* Have a clinical diagnosis of moderate to severe chronic plaque psoriasis and be a candidate for treatment with Raptiva®.
* Are being treated or are initiating treatment with Raptiva® at time of study enrolment in accordance with the Canadian Product Monograph indication and recommendations.
* Be able to provide written informed consent.
* Agreement to participate in the study, and to disclose any medical events to the Investigator.
* The subject must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

* Any contra-indication to Raptiva® according to the Canadian Product Monograph.
* Any simultaneous participation in another clinical evaluation trial for psoriasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting Raptiva® (efalizumab) treated patients with moderate to severe chronic plaque psoriasis and meeting the inclusion/exclusion criteria specified will be eligible for participation in this study. Subjects will be enrolled from the Raptiva®-treated clinical patient pool at the participating Canadian investigator site.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
All serious and unexpected AEs | During the course of the study

SECONDARY OUTCOMES:
Investigator assessed: static Physician's Global Assessment (sPGA). Patient assessed: Dermatology Life Quality Index (DLQI) | During the course of the study, there are no pre-defined scheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Horia Ijacu, MD, Study Director — EMD Canada Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Medical Information - Canada, Mississauga, Ontario, Canada